CLINICAL TRIAL: NCT06022380
Title: COHERE - Core Outcome Set for Head, Neck and Respiratory Disease in Mucopolysaccharidosis II
Brief Title: Core Outcome Set for Head, Neck and Respiratory Disease in Mucopolysaccharidosis II
Acronym: COHERE
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B00446 - COHERE; 261752 (Other: IRAS ID)
Record Dates: First submitted 2023-08-24; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Mucopolysaccharidosis Type II
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Round 1: Participants will be asked to score each outcome domain on a 9 point scale proposed by the GRADE group [http://www.gradeworkinggroup.org], in which 1 to 3 signifies an outcome of 'limited importance', 4 to 6 'important but not critical', and 7 to 9 'critical'. Round 1 will also provide participants with the opportunity to add further outcomes which they think may be important. Any suggested outcomes deemed to represent a new outcome domain by the study group (following discussion within study advisory group and a majority decision) will be added to the list for consideration in round two. Round 1 will last for approximately 2 months.
- Round 2: All items (in addition to further new outcome domains identified by participants in round 1) will be carried forward for consideration in round 2. Descriptive statistics (graphs) will be used to summarize the scores from round 1 and presented to participants. Participants will see the results of their individual score for each outcome in addition to the median score of each stakeholder group. The rationale for showing participants the scores from other groups is that it may improve consensus between the stakeholder groups. In addition, by carrying all items forward from round 1, it may be possible to identify changes in scoring patterns as a result of viewing other scores. Participants will be asked to score all items once again using the 9-point scale. Round 2 will last for approximately 2 month

SUMMARY:
The Mucopolysaccharidoses (MPS) are a family of genetic metabolic disorders, caused by specific enzyme deficiencies which result in accumulation of partially degraded glycosaminoglycans (GAGs) within various tissues. As GAGs are common in the body a number of different organ systems can be affected. Involvement of the upper and lower respiratory tract in MPS Type II results in significant airway compromise, with progressive airway obstruction being responsible for a significant proportion of the morbidity and mortality associated with this condition. Hearing loss is a universal finding in MPS, with a third of patients suffering with severe profound hearing loss. There is an unmet need for strong clinical evidence to guide treatment of head, neck and respiratory disease in MPS disorders. A Core Outcome Set (COS) describes the minimum outcome data that should be measured in a clinical study for a particular condition. The lack of an agreed COS for MPS II in general, and specifically head, neck and respiratory disease, makes comparison between studies difficult. There is also a lack of information detailing patient and parent perspectives on the MPS disorders. The ideal COS for head, neck and respiratory disease associated with MPS II would combine both patient/parent and clinician opinion and could be used in the design of all subsequent clinical studies. Following literature review the investigators have created a list of outcomes previously reported for qualitative and quantitative studies investigating head, neck and respiratory disease in MPS II. For the proposed research the investigators will seek opinions of patients, parents, clinicians and scientists to rate these outcomes via the Delphi method. Outcomes scored highest by patients, parents, clinicians and scientists will form a COS for head, neck and respiratory disease in MPS II. The development of a COS can help limit variability outcomes in studies investigating different interventions in MPS II.

ELIGIBILITY:
Inclusion criteria:

* Confirmed MPS II diagnosis.
* Aged between 12 and 25 years old.
* Parents/ main care givers of child with MPS Type II.
* Adults aged 18 or over.
* Clinicians responsible for direct care and management of at least 2 pediatric MPS Type II patients in the last 12 months.
* Scientists who have worked with MPS Type II within the last 5 years

Exclusion criteria:

* Unconfirmed MPS Type II diagnosis.
* Aged below 12 and above 25 years old.
* Not directly involved in a day to day care.
* Clinicians who only occasionally look after pediatric MPS Type II patients.
* Scientists who have not worked with MPS Type II within the last 5 years

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients and parents, clinicians and scientists
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
What are the most important outcomes that should be measured in trials examining ENT and respiratory disease in MPS Type II populations, aged 0-11 and 12-25 years old? | 8 months
  Step 1. A systematic review of the literature and clinical trials registries (including the Hunter Outcome Survey) was undertaken to identify a comprehensive list of head, neck and respiratory disease outcomes reported in literature and trials of MPS Type II population. Additionally, qualitative research investigated perspectives of patients with MPS Type II.
  Step 2. A Delphi survey of 3 key stakeholder groups (Patients (only for COS for the age group 12-25 years old), parents/ care givers, MPS Type II healthcare professionals), will be undertaken to try to achieve consensus about the outcomes to include in a COS.
  Step 3, This will be followed by a consensus meeting of key stakeholders to ratify the COS.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Lancashire, United Kingdom